CLINICAL TRIAL: NCT06315608
Title: An Open-Label, Proof of Concept Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of MRG-001 in Patients With Amyotrophic Lateral Sclerosis
Brief Title: MRG-001 in Patients With Amyotrophic Lateral Sclerosis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedRegen LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG24ALS
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Amyotrophic Lateral Sclerosis; Lou Gehrig Disease; Motor Neuron Disease; Motor Neuron Atrophy
Keywords: MRG-001; Stem Cells; Regulatory T-cells; Fixed-Dose Combination
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MRG-001 (0.01 mL/kg) (Experimental): MRG-001 will be subcutaneously administered at 0.01 mL/kg 3 times per week every other day for two weeks per month (Day 0, 2, 4, 7, 9, 11). This cycle will be repeated 3 months in total.
  Interventions: Drug: MRG-001

INTERVENTIONS:
Drug: MRG-001 — MRG-001 is a clear liquid solution for subcutaneous injection

SUMMARY:
The proposed study is an Open-Label, Single-Dose Study to Assess the Safety, and Pharmacodynamics (PD) signals of MRG-001 in Patients with Amyotrophic Lateral Sclerosis (ALS). MRG-001 will be administered subcutaneously 3 times per week for 2 weeks. This cycle will be repeated for 3 months. In total, patients are expected to receive 18 injections over the span of 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent (either from patient or patient's legally acceptable representative and complying with study procedures, in the PI's opinion.
* Male or female patients between 18-75 years.
* Sporadic or familial ALS diagnosed as clinically possible, probable, lab-supported probable, or definite ALS defined by revised El Escorial criteria.
* Time since onset of weakness due to ALS ≤ 48 months at the time of the Screening Visit
* Vital Capacity ≥ 50% of predicted capacity for age, height, and sex at the time of the Screening Visit measured by Slow Vital Capacity (SVC), or Forced Vital Capacity (FVC).
* Patients must either not take Riluzole or be on a stable dose of Riluzole for ≥ 30 days prior to the Master Protocol Screening Visit. Riluzole-naïve participants are permitted in the study.
* Participants must either not take Edaravone or have completed at least one cycle of edaravone prior to the Master Protocol Screening Visit. Edaravone-naïve participants are permitted in the study.
* Participants must either not take Relyvrio (AMX0035) or be on a stable dose of Relyvrio for ≥ 30 days prior to the Master Protocol Screening Visit. Relyvrio-naïve participants are permitted in the study.
* Women of child-bearing potential (defined as females who are not surgically sterile or who are not over the age of 52 and amenorrhoeic for at least 12 months) must utilize appropriate birth control throughout the study duration.
* Male patients must agree to use a medically acceptable method of contraception /birth control throughout the study duration.

Exclusion Criteria:

* Subjects who meet one or more of the following criteria will not be considered eligible to participate in the clinical study:
* Participation in another interventional clinical trial (drug or device) within 30 days of Screening and at any time during the study.
* Significant pre-existing organ dysfunction prior to randomization:
* Lung: Receiving supplemental home oxygen therapy at baseline for pre-existing medical condition (other than COVID-19), as documented in medical record.
* Heart: Pre-existing congestive heart failure defined as an ejection fraction <20% as documented in the medical record. Clinically significant ventricular arrhythmias (ventricular tachycardia, ventricular fibrillation), unstable angina, myocardial infarction (past 3 months), heart and coronary vessel surgery (past 3 months), significant valvular heart disease, uncontrolled arterial hypertension with systolic blood pressure >180 mm Hg and diastolic blood pressure >110 mm Hg.
* Renal: End-stage renal disease requiring renal replacement therapy or creatinine clearance <50 mL/min.
* Hematologic: Baseline platelet count <30,000/mm3 or hemoglobin levels <6.0 g/dL.
* Neurological: Stage ≥3 hepatic encephalopathy by West Haven criteria.
* History of splenectomy or splenomegaly (spleen weighing > 750 g).
* Active cancer or history of cancer, except for the following: basal cell carcinoma or successfully treated squamous cell carcinoma of the skin, cervical carcinoma in situ, prostatic carcinoma in situ, or other malignancies curatively treated and with no evidence of disease recurrence for at least 3 years.
* Presence of unstable psychiatric disease, cognitive impairment, dementia or substance abuse that would impair ability of the participant to provide informed consent, in the SI's opinion.
* Exposure at any time to any gene therapies under investigation for the treatment of ALS (off-label use or investigational) including tofersen (Qalsody).
* History of splenectomy or splenomegaly (spleen weighing >750 g).
* Co-infection with human immunodeficiency virus (HIV).
* History of organ or bone marrow transplantation, other than a corneal transplant.

or recent (within 3 months) chronic use of immunosuppressive drugs (tacrolimus, mycofenolate mofetil, cyclosporine, rapamycine, hydrochloroquine, azathiopurine, methotrexate), e.g., biologicals, JAK1/2 inhibitors, interferons, interleukins or (prednisone or related corticosteroids are allowed).

* Hypersensitivity to either of the components of MRG-001.
* If female, known pregnancy, or has a positive serum pregnancy test, or lactating/breastfeeding.
* Underlying diseases that, in the opinion of the site investigator, might be complicated or exacerbated by proposed treatments or might confound assessment of study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Treatment-Emergent Adverse Events | 3 Months
  Assess the safety and tolerability of MRG-001 in patients with Amyotrophic Lateral Sclerosis (ALS) as determined by the absence of serious adverse events (SAE)

SECONDARY OUTCOMES:
Stem Cell Mobilization | 24 hours
  The absolute change in numbers of CD34+ hematopoetic stem cells as measured by flow cytometry
Regulatory T-cell Mobilization | 24 hours
  The absolute change in numbers of FOXP3+ regulatory T-cells as measured by flow cytometry
Change in Disease Progression | 3 Months
  Change in disease severity over time as measured by the ALS Functional Rating Scale-Revised (ALSFRS-R) at Baseline, 1, 2 and 3 months. Each type of function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function. Positive data means the reversal of ALS disease, negative data means disease progression, zero means stabilization of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Ali R Ahmadi, MD PhD, Study Director — MedRegen LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahmadi AR, Atiee G, Chapman B, Reynolds L, Sun J, Cameron AM, Wesson RN, Burdick JF, Sun Z. A phase I, first-in-human study to evaluate the safety and tolerability, pharmacokinetics, and pharmacodynamics of MRG-001 in healthy subjects. Cell Rep Med. 2023 Sep 19;4(9):101169. doi: 10.1016/j.xcrm.2023.101169. Epub 2023 Aug 25. PMID 37633275
- See also: Company Profile — http://medregenco.com